CLINICAL TRIAL: NCT03877185
Title: A New Revolutionary 3-Injection- Protocol in Infertile Women With a Single Long Acting GnRH Antagonist in the Luteal Phase, a Bolus Gonadotropin Injection in the Early Follicular Phase and a Single Triggering Dose.
Brief Title: A New Revolutionary 3-Injection- Protocol in Infertile Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assisting Nature (Other)
Responsible Party: Principal Investigator, Papanikolaou Evaggelos, Papanikolaou Evaggelos, MD, PhD, Fertility Specialist, Scientific Director at Assisting Nature IVF Clinic, Assisting Nature
Other Study IDs: 3-Injection-Protocol-AN008
Record Dates: First submitted 2019-03-14; First posted 2019-03-15 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Infertility, Female
Keywords: IVF; infertility; long antagonist; long acting gonadotropin; corifollitropin alfa; ovarian stimulation
MeSH Terms: conditions — Infertility, Female; Infertility | interventions — Pregnancy Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 3-Injection-Protocol Group: Women in group A (3-Injection-Protocol Group) receive a bolus late luteal dose of Degarelix, a new long acting GnRH antagonist, a sole Elonva injection in the early follicular phase followed by the administration of a single dose of triggering agent (GnRH agonist or hCG a, according to the individual response).
  Interventions: Diagnostic Test: Live birth rate
- Multiple-Injection- Protocol Group: Women assigned to group B (Multiple- Injection- Protocol Group) are administered a single dose of Elonva (corifollitropin alfa) in the early follicular phase followed by daily GnRH antagonist doses, either fixed on day 6 of the stimulation cycle, or when 2 or 3 follicles over 12-14 mm are present. Ovulation triggering is the same as in group A, with either GnRH agonist or hCG a, accordingly.
  Interventions: Diagnostic Test: Live birth rate

INTERVENTIONS:
Diagnostic Test: Live birth rate — Live Birth Rate and Blastulation Rate according to the protocol of COS
  Other Names: Blastulation rate

SUMMARY:
This is a prospective randomised study of the evaluation of the clinical IVF results after following a new revolutionary 3-Injection- Protocol for controlled ovarian stimulation in infertile women.

DETAILED DESCRIPTION:
A randomized prospective study focusing on infertile women undergoing ovarian stimulation for IVF, using Elonva (corifollitropin alfa) as part of two different stimulation protocols.

Women assigned to Protocol A receive a bolus late luteal dose of Degarelix, a new long acting GnRH antagonist, a sole Elonva injection in the evening of day 3 of the cycle, followed by the administration of a single dose of triggering agent (GnRH agonist or hCG a, according to the individual response).

Women assigned to Protocol B are administered a single dose of Elonva (corifollitropin alfa) on day 2 of the cycle, followed by daily GnRH antagonist doses, fixed on day 7 of the cycle. Ovulation triggering is the same as in group A, with either GnRH agonist or hCG a, accordingly.

Live Birth Rates are estimated for both groups of patients. The number of the formed blastocysts in each group is measured, as well.

ELIGIBILITY:
Inclusion Criteria:

* primary infertility
* age 22-39 years;
* body mass index (BMI) 18-29kg/m2;
* regular menstrual cycle of 26-35 days,
* presumed to be ovulatory;
* early follicular- phase serum concentration of FSH within normal limits (1-12 IU/l).

Exclusion Criteria:

* women with diabetes and other metabolic disease
* women with heart disease, QT prolongation, heart failure
* elevated liver enzymes, liver failure, hepatitis
* women with inflammatory or autoimmune disease
* abnormal karyotype
* polycystic ovarian syndrome
* endometriosis stage III/IV

Ages: 22 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women aged 22- 39, faced with infertility issues, meeting the above inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Live birth rate according to stimulation protocol | Up to 38 weeks after embryo transfer
  Live birth rate according to stimulation protocol

SECONDARY OUTCOMES:
Blastulation rate according to stimulation protocol | Up to 6 days post oocyte retrieval
  Blastulation rate according to stimulation protocol

CONTACTS AND LOCATIONS:
Overall Officials: Evaggelos Papanikolaou, MD,PhD, Principal Investigator — Assisting Nature; Robert Najdecki, MD,PhD, Principal Investigator — Assisting Nature
Locations (1):
- Assisting Nature, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided